CLINICAL TRIAL: NCT04542538
Title: The Impact of Premorbid Illnesses on the Risk of ICU Admission and Short-term Outcome
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Center for Clinical Research Dalarna, Sweden (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1257-2830
Record Dates: First submitted 2020-08-21; First posted 2020-09-09 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Sepsis; Corona Virus Infection; ARDS, Human
MeSH Terms: conditions — Sepsis; Coronavirus Infections; Respiratory Distress Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 critical care patients: All patients who have received intensive care with COVID-19 in Sweden until May 27, 2020. Patients are identified in the Swedish Intensive care registry, to which all Swedish intensive care units (ICU) are reporting all intensive care patients.
  Interventions: Other: No intervention, observational study
- Sepsis critical care patients: All patients who have received intensive care with severe sepsis or septic shock in Sweden between 2011 and 2016. Patients are identified in the Swedish Intensive care registry, to which all Swedish intensive care units (ICU) are reporting all intensive care patients.
  Interventions: Other: No intervention, observational study
- ARDS critical care patients: All patients who have received intensive care with ARDS in Sweden between 2011 and 2016. Patients are identified in the Swedish Intensive care registry, to which all Swedish intensive care units (ICU) are reporting all intensive care patients.
  Interventions: Other: No intervention, observational study

INTERVENTIONS:
Other: No intervention, observational study

SUMMARY:
The Corona virus disease 2019 (COVID-19) pandemic is currently involving all parts of the world. Several risk factors for critical illness and death from the disease have been proposed. However, it is still unclear if the observed associations between different comorbidities and chronic medications and severe COVID-19 disease and mortality is different from associations between the same factors and other severe diseases requiring intensive care unit (ICU) -care. This is important since some of the observed risk factors are very common in the aged who, by age alone, are more prone to a more severe course of any disease. By combining several registries, this study will compare, on several comorbidities such as hypertension and diabetes , the first 2000 cases of COVID-19 patients receiving critical care in Sweden to a Swedish sepsis-cohort and a Swedish adult respiratory distress syndrome (ARDS) -cohort.

DETAILED DESCRIPTION:
The Corona virus disease 2019 (COVID-19) pandemic is currently involving all parts of the world. Several risk factors for critical illness and death from the disease have been proposed. However, it is still unclear if the observed associations between different comorbidities and chronic medications and severe COVID-19 disease and mortality is different from associations between the same factors and other severe diseases requiring ICU-care. This is important since some of the observed risk factors are very common in the aged who, by age alone, are more prone to a more severe course of any disease. By combining several registries, this study will compare, on several comorbidities such as hypertension and diabetes , the first 2000 cases of COVID-19 patients receiving critical care in Sweden to a Swedish sepsis-cohort and a Swedish ARDS-cohort.

ELIGIBILITY:
Inclusion Criteria:

° Individual registered in the Swedish intensive care registry (SIR) with COVID-19 Before 27 May 2020.

or

* Individual registered in the SIR with Severe sepsis or septic chock 2011-2016. or
* Individual registered in the SIR with ARDS 2011-2016.

Exclusion Criteria:

* Age below 18 years
* Individual registered in the Swedish intensive care registry without a personal identification number

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The SIR is a registry to which all Swedish intensive care units are reporting all intensive care patients. The SIR has a specific part to wich all COVID-19 related intensive care eposodes are reported. All patients, approximally 2000, who have at least one COVID-19 listing in the SIRI will be included, as cases. Two historical control populations are extracted from the SIR between 2011 and 2016. One population with all patients having had severe sepsis and one with all patients having had ARDS during ICU care.
  We already have recieved all data on the studypopulation and the Control populations but will not set up the database or perform any analyses until this registration is be public.
Sampling Method: Probability Sample
Enrollment: 9905 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
Risk factors of ICU care COVID-19/Sepsis | Five years preceding ICU admission to ICU admission
  In a binary logistics model with the outcome Sepsis or COVID-19 the OR for several comorbidities are determined.
Risk factors of ICU care COVID-19/ARDS | Five years preceding ICU admission to ICU admission
  In a binary logistics model with the outcome ARDS or COVID-19 the OR for several comorbidities are determined.
Risk factors of ICU mortality COVID-19/Sepsis | Five years preceding ICU admission to ICU discharge
  In a Cox proportional hazards model with the outcome ICU-mortality the hazard ratio (HR) for the interaction between several comorbidities and a binary variable COVID-19/Sepsis are determined.
Risk factors of ICU mortality COVID-19/ARDS | Five years preceding ICU admission to ICU discharge
  In a Cox proportional hazards model with the outcome ICU-mortality the HR for the interaction between several comorbidities and a binary variable COVID-19/ARDS are determined.

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Lipcsey, PhD, Principal Investigator — Uppsala University
Locations (1):
- Björn Ahlström, Falun, Sweden

IPD SHARING:
Plan to Share IPD: No